CLINICAL TRIAL: NCT06312761
Title: Single-Dose Pharmacokinetics of Oral Testosterone Undecanoate With and Without Concomitant Inhibition of UGT2B17 With Oral Curcumin in Normal Men With Experimental Hypogonadism
Brief Title: Single-Dose Pharmacokinetics of Oral Testosterone Undecanoate With and Without Concomitant Inhibition of UGT2B17
Acronym: OralT12
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Washington State University (Other)
Responsible Party: Principal Investigator, John Amory, Professor, DOM - General Internal Medicine, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Oral T-12
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Hypogonadism, Male
Keywords: Oral Testosterone undecanoate; Hypogonadism; Curcumin; Testosterone replacement therapy
MeSH Terms: conditions — Eunuchism; Hypogonadism | interventions — relugolix; Curcumin; testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 Oral testosterone undecanoate without Curcumin (Experimental): Oral testosterone undecanoate 237 mg Day 2
  Interventions: Drug: Testosterone Undecanoate 237 MG Oral Capsule
- Arm 2 Oral testosterone undecanoate with Curcumin (Experimental): Oral testosterone undecanoate 237 mg & Curcumin 630 mg Day 3
  Interventions: Dietary Supplement: Curcumin; Drug: Testosterone Undecanoate 237 MG Oral Capsule
- Relugolix 120 mg single dose (Other): All subjects will received Relugoliz on Day 1
  Interventions: Drug: Relugolix 120Mg Tab

INTERVENTIONS:
Drug: Relugolix 120Mg Tab — Relugolix 120 mg single dose - All subjects
  Arms: Relugolix 120 mg single dose
Dietary Supplement: Curcumin — Curcumin 630 mg single dose
  Arms: Arm 2 Oral testosterone undecanoate with Curcumin
Drug: Testosterone Undecanoate 237 MG Oral Capsule — Testosterone Undecanoate 237 MG Oral Capsule
  Arms: Arm 1 Oral testosterone undecanoate without Curcumin; Arm 2 Oral testosterone undecanoate with Curcumin

SUMMARY:
This study will be performed in normal men whose endogenous testosterone production has been temporarily suppressed by the administration of a single dose of 120 mg of the oral GnRH antagonist Relugolix, which is approved for the treatment of prostate cancer, and can suppress endogenous testosterone biosynthesis for 48-72 hours after a single dose.

DETAILED DESCRIPTION:
The study will have three phases: a screening period, a 3-day drug exposure period, and a one-month recovery period (see Table 1, Experimental Design).

Screening Visit: At screening, study investigators will consent subjects, perform an interview and physical examination; blood samples for measurement of hormones (T,

DHT, Estradiol (E2), FSH and LH), routine hematology, chemistry and hepatic function and a DNA sample for UGT2B17 genotype will be obtained from the buccal mucosa and a spot urine specimen obtained for a testosterone glucuronide/androsterone glucuronide ratio (a marker of endogenous UGT2B17 activity). No drugs will be administered in the screening period. The screening visit should take approximately 60 minutes.

Day 1 (15-minute visit): Blood pressure and heart rate will be measured prior to the administration of Relugolix 120 mg orally on an empty stomach.

Day 2 (9 hour stay): Placement of IV and dosing of Testosterone Undecanoate 237 mg once with two ensures. The first dose of oral testosterone will be administered at 0900 (+/- 30 minutes) in the morning with two Ensures. After drug administration, subjects will have 10 ccs of blood drawn for the measurement of serum testosterone for the measurement of testosterone Predose, 0.5, 1, 1.5 2, 3, 4, 6, and 8 hours after the morning dose and will have the iv removed.

Day 3 (9 hour stay): Placement of IV and dosing of Testosterone Undecanoate 237 mg once with two Ensures and 630 mg of oral Curcumin. The second dose of oral testosterone will be administered at 0900 (+/- 30 minutes) in the morning. After drug administration, subjects will have 10 ccs of blood drawn for the measurement of serum testosterone for the measurement of testosterone Predose, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours after the morning dose and will have the iv removed.

Day 4 (15-minute visit): Subjects will come into the clinic at 0900 for a 24-hour blood draw and adverse effect assessment.

Day 28-42 (30-minute visit): Subjects will undergo a final assessment (physical examination, vitals and weight measurements and blood draw) on day 28-42. We will confirm at the follow-up visit that there has been recovery from Relugolix-induced hypogonadism (i.e., testosterone levels have returned to within 25% of baseline). If a subject has not recovered by this visit, he will be reassessed at 2-week intervals until recovery is documented. The total amount of blood drawn over the study protocol will not exceed 500 mL per subject.

ELIGIBILITY:
Inclusion Criteria:

* 1. healthy male between 18 and 55 years of age
* 2. agrees to not participate in another drug research study for the duration of this study
* 3. agrees to not donate blood during the study
* 4. subject provided written (personally signed and dated) informed consent before completing any study-related procedures
* 5. subject able and willing to comply with the protocol
* 6. subject able and willing to not take medications other than the study drug for the duration of the study

Exclusion Criteria:

* 1. subject has poor general health, determined by medical history or physical exam
* 2. subject have an abnormal evaluation on screening exam (consisting of serum chemistry, hematology and baseline hormone levels)
* 3. subject have a known history or current use of alcohol drug or steroid abuse and/or the use of more than 3 alcoholic beverages per day
* 4. History of current testosterone use
* 5. History of testicular disease or severe testicular trauma
* 6. History of major psychiatric disorder
* 7. subject participated in a hormonal drug study within the past month
* 8. Subject or his partner(s) NOT willing to use an accepted method of contraception during the study
* 9. History of Bleeding disorders or current use of anti-coagulants

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
average serum testosterone after dosing on day 2 | 24 hour period (between dosing at beginning of day 2 and end of day 2)
average serum testosterone after dosing on day 3 | 24 hour period (between dosing at beginning of day 3 and end of day 3)
Maximum concentration | Cmax during 24 hour period (between dosing at beginning of day 2 and 3 and end of day 2 or day 3)
time to maximum concentration | T max during 24 hour period (between dosing at beginning of day 2 and 3 and end of day 2 or day 3)
area-under-the curve | 24 hour period (between dosing at beginning of day 2 and 3 and end of day 2 or day 3)
elimination phase half-life | 24 hour period (between dosing at beginning of day 2 and 3 and end of day 2 or day 3)

CONTACTS AND LOCATIONS:
Overall Officials: John Amory, MD, Principal Investigator — University of Washington

REFERENCES:
- [Background] Katznelson L, Finkelstein JS, Schoenfeld DA, Rosenthal DI, Anderson EJ, Klibanski A. Increase in bone density and lean body mass during testosterone administration in men with acquired hypogonadism. J Clin Endocrinol Metab. 1996 Dec;81(12):4358-65. doi: 10.1210/jcem.81.12.8954042.
- [Background] Behre HM, Kliesch S, Leifke E, Link TM, Nieschlag E. Long-term effect of testosterone therapy on bone mineral density in hypogonadal men. J Clin Endocrinol Metab. 1997 Aug;82(8):2386-90. doi: 10.1210/jcem.82.8.4163. PMID 9253305
- [Background] Bhasin S, Bremner WJ. Clinical review 85: Emerging issues in androgen replacement therapy. J Clin Endocrinol Metab. 1997 Jan;82(1):3-8. doi: 10.1210/jcem.82.1.3640. No abstract available. PMID 8989221
- [Background] Plymate SR "Male Hypogonadism" in Principles and Practice of Endocrinology and Metabolism (3rd. Ed). Ed. Kenneth Becker, pp:1125-1150
- [Background] Wang C, Alexander G, Berman N, Salehian B, Davidson T, McDonald V, Steiner B, Hull L, Callegari C, Swerdloff RS. Testosterone replacement therapy improves mood in hypogonadal men--a clinical research center study. J Clin Endocrinol Metab. 1996 Oct;81(10):3578-83. doi: 10.1210/jcem.81.10.8855804.
- [Background] Wang C, Swerdloff RS. Testosterone Replacement Therapy in Hypogonadal Men. Endocrinol Metab Clin North Am. 2022 Mar;51(1):77-98. doi: 10.1016/j.ecl.2021.11.005. Epub 2022 Feb 8. PMID 35216722
- [Background] Kelch RP, Jenner MR, Weinstein R, Kaplan SL, Grumbach MM. Estradiol and testosterone secretion by human, simian, and canine testes, in males with hypogonadism and in male pseudohermaphrodites with the feminizing testes syndrome. J Clin Invest. 1972 Apr;51(4):824-30. doi: 10.1172/JCI106877. PMID 4259253
- [Background] Weinstein RL, Kelch RP, Jenner MR, Kaplan SL, Grumbach MM. Secretion of unconjugated androgens and estrogens by the normal and abnormal human testis before and after human chorionic gonadotropin. J Clin Invest. 1974 Jan;53(1):1-6. doi: 10.1172/JCI107526. PMID 4271572
- [Background] Bagatell CJ, Bremner WJ. Androgens in men--uses and abuses. N Engl J Med. 1996 Mar 14;334(11):707-14. doi: 10.1056/NEJM199603143341107. No abstract available. PMID 8594431
- [Background] Fossa SD, Opjordsmoen S, Haug E. Androgen replacement and quality of life in patients treated for bilateral testicular cancer. Eur J Cancer. 1999 Aug;35(8):1220-5. doi: 10.1016/s0959-8049(99)00123-9. PMID 10615233
- [Background] Amory JK, Matsumoto AM. The therapeutic potential of testosterone patches. Expert Opin Investig Drugs. 1998 Dec;7(12):1977-85. doi: 10.1517/13543784.7.12.1977. PMID 15991940
- [Background] Swerdloff RS, Wang C, Cunningham G, Dobs A, Iranmanesh A, Matsumoto AM, Snyder PJ, Weber T, Longstreth J, Berman N. Long-term pharmacokinetics of transdermal testosterone gel in hypogonadal men. J Clin Endocrinol Metab. 2000 Dec;85(12):4500-10. doi: 10.1210/jcem.85.12.7045. PMID 11134099
- [Background] de Ronde W. Hyperandrogenism after transfer of topical testosterone gel: case report and review of published and unpublished studies. Hum Reprod. 2009 Feb;24(2):425-8. doi: 10.1093/humrep/den372. Epub 2008 Oct 23. PMID 18948313
- [Background] Swerdloff RS, Dudley RE. A new oral testosterone undecanoate therapy comes of age for the treatment of hypogonadal men. Ther Adv Urol. 2020 Jun 30;12:1756287220937232. doi: 10.1177/1756287220937232. eCollection 2020 Jan-Dec. PMID 32655691
- [Background] Bhatt DK, Basit A, Zhang H, Gaedigk A, Lee SB, Claw KG, Mehrotra A, Chaudhry AS, Pearce RE, Gaedigk R, Broeckel U, Thornton TA, Nickerson DA, Schuetz EG, Amory JK, Leeder JS, Prasad B. Hepatic Abundance and Activity of Androgen- and Drug-Metabolizing Enzyme UGT2B17 Are Associated with Genotype, Age, and Sex. Drug Metab Dispos. 2018 Jun;46(6):888-896. doi: 10.1124/dmd.118.080952. Epub 2018 Mar 30. PMID 29602798
- [Background] Basit A, Amory JK, Mettu VS, Li CY, Heyward S, Jariwala PB, Redinbo MR, Prasad B. Relevance of Human Aldoketoreductases and Microbial beta-Glucuronidases in Testosterone Disposition. Drug Metab Dispos. 2023 Apr;51(4):427-435. doi: 10.1124/dmd.122.000975. Epub 2023 Jan 9. PMID 36623880
- [Background] MacLean DB, Shi H, Faessel HM, Saad F. Medical Castration Using the Investigational Oral GnRH Antagonist TAK-385 (Relugolix): Phase 1 Study in Healthy Males. J Clin Endocrinol Metab. 2015 Dec;100(12):4579-87. doi: 10.1210/jc.2015-2770. Epub 2015 Oct 26. PMID 26502357